CLINICAL TRIAL: NCT01759277
Title: Femoral Versus Adductor Canal Continuous Peripheral Nerve Blocks for Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Summit Medical Products, Inc. (Unknown); Teleflex (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adductor Canal vs Femoral
Record Dates: First submitted 2012-12-21; First posted 2013-01-03 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain Following Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Femoral perineural local anesthetic infusion
  Interventions: Drug: Control: Femoral perineural local anesthetic infusion
- Experimental (Experimental): Adductor canal perineural local anesthetic infusion
  Interventions: Drug: Experimental: Adductor Canal perineural local anesthetic infusion

INTERVENTIONS:
Drug: Control: Femoral perineural local anesthetic infusion — The control group will receive a femoral nerve block and postoperative ropivacaine 0.2% infusion
  Arms: Control
Drug: Experimental: Adductor Canal perineural local anesthetic infusion — The control group will receive an adductor canal nerve block and postoperative ropivacaine 0.2% infusion
  Arms: Experimental

SUMMARY:
Patients typically experience moderate-to-severe pain following knee arthroplasty that is usually treated with a combination of oral and intravenous analgesics and enhanced by continuous peripheral nerve blocks. There are currently two locations to place a perineural catheter to provide analgesia following knee arthroplasty: a femoral nerve catheter and an adductor canal catheter. Both have been demonstrated to be effective following knee arthroplasty. However, it remains unknown if one location is superior to the other; or, more accurately, what the relative benefits are to each technique.

While femoral CPNB has many benefits, one of the challenges of using this technique is that there is a decrease in quadriceps muscle strength which can be a limiting factor for rehabilitation. In contrast, the adductor canal catheter affects only the vastus medialis. This block may lessen block-induced quadriceps weakness following knee arthroplasty compared with a femoral infusion.

The investigators hypothesize that compared with femoral perineural local anesthetic infusion, an adductor canal infusion is associated with a shorter time until four discharge criteria are met: (1) adequate analgesia; (2) independence from intravenous analgesics; (3) ability to ambulate 30 m; and (4) ability to stand, walk 3 m, and return to a sitting position without another's assistance.

DETAILED DESCRIPTION:
Of importance: The primary investigation involves 80 evaluable subjects (with primary endpoint data) having tri-compartment knee arthroplasty. In addition, the investigators will enroll up to 70 subjects having uni-compartment knee arthroplasty as a pilot study in preparation for a subsequent larger, definitive trial. These two groups will not be analyzed together--they represent two distinct studies: one a definitive RCT for tri-compartment knee arthroplasty; and, one a pilot study for uni-compartment knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. primary, unilateral knee arthroplasty
2. age ≥ 18 years
3. postoperative analgesic plan includes perineural local anesthetic infusion of 48-72 hours

Exclusion Criteria:

1. morbid obesity as defined by a body mass index >40 (BMI=weight in kg/ [height in meters]
2. chronic, high-dose opioid use (greater than 20mg oxycodone-equivalent opioid use daily within the 2 weeks prior to surgery and duration of use >4 weeks)
3. history of opioid abuse
4. allergy to study medications
5. known renal insufficiency (creatinine > 1.5 mg/dL)
6. pregnancy
7. incarceration
8. any known neuro-muscular deficit of the ipsilateral femoral nerve, obturator nerve and/or quadriceps muscle (including diabetic peripheral neuropathy); and inability to ambulate 30 m preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego
Locations (1):
- University of California San Diego Medical Centers, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Ilfeld BM, Loland VJ, Sandhu NS, Suresh PJ, Bishop MJ, Donohue MC, Ferguson EJ, Madison SJ. Continuous femoral nerve blocks: the impact of catheter tip location relative to the femoral nerve (anterior versus posterior) on quadriceps weakness and cutaneous sensory block. Anesth Analg. 2012 Sep;115(3):721-7. doi: 10.1213/ANE.0b013e318261f326. Epub 2012 Jun 28. PMID 22745116
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Background] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- [Background] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Femoral perineural local anesthetic infusion
  Active comparator: Control: Femoral perineural local anesthetic infusion: The control group will receive a femoral nerve catheter and block under ultrasound guidance with the final position of catheter posterior to the femoral nerve and lateral to the femoral artery. Normal saline up to 10ml will be injected if necessary for hydro-dissection via the needle. The catheter will then be threaded 3-5cm past the needle tip and its location will be confirmed by a 30ml bolus of lidocaine 2% via the catheter under ultrasound visualization. The control group will receive a standardized general anesthetic with inhaled volatile anesthesia in nitrous oxide and oxygen or bupivacaine spinal anesthetic.
- Experimental: Adductor canal perineural local anesthetic infusion
  Experimental: Adductor Canal perineural local anesthetic infusion: The experimental group will receive an adductor canal catheter and block under ultrasound guidance with the final position of catheter between the femoral artery and nerve. Normal saline up to 10ml will be injected if necessary for hydro-dissection via the needle. The catheter will then be threaded 3-5cm past the needle tip and its location will be confirmed by a 30ml bolus of lidocaine 2% via the catheter under ultrasound visualization. The control group will receive a standardized general anesthetic with inhaled volatile anesthesia in nitrous oxide and oxygen or bupivacaine spinal anesthetic.
Period: Overall Study
Arm/Group | Control | Experimental
Started | 41 | 39
Completed | 41 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7) | 67 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 14 | 16 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 168 (10) | 169 (11) | 169 (11)
Weight [Mean (Standard Deviation); unit: kg] | 84 (16) | 87 (16) | 86 (17)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29 (5) | 30 (5) | 30 (5)

OUTCOME MEASURES:

1. Primary Outcome: Hours Until Discharge Readiness
Description: Discharge readiness is the number of hours until meeting the following 4 criteria: (1) adequate analgesia (defined as pain less than 4 on a NRS of 0-10); (2) independence from intravenous analgesics; (3) ability to ambulate 30 m and (4) ability to stand, walk 3 m, and return to a sitting position without another's assistance.
Time Frame: 7 postoperative days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control | Experimental
Number analyzed (Participants) | 41 | 39
hours | 61 [49 to 69] | 55 [42 to 63]

2. Secondary Outcome: Time to Adequate Analgesia
Description: The time in hours until adequate analgesia is defined as pain less than 4 on a Numeric Rating Scale of 0-10, with 0=no pain and 10=worst imaginable pain
Time Frame: First 7 postoperative days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Control | Experimental
Number analyzed (Participants) | 41 | 39
Hours | 61.6 (20.2) | 61.0 (19.3)

3. Secondary Outcome: Time Until Independence From Intravenous Analgesics of at Least 12 Hours
Description: The time in hours until no intravenous analgesics were required for at least 12 hours (without future intravenous use during admission)
Time Frame: First 7 postoperative days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Control | Experimental
Number analyzed (Participants) | 41 | 39
Hours | 46.1 (20.1) | 47.5 (22.7)

4. Secondary Outcome: Time Until Timed Up and Go Test Achieved
Description: The timed-up-and-go (TUG) test measures the ability and speed of standing from a sitting position, walking 3 meters and returning to the original seated position independent from the assistance of healthcare personnel. This variable measured the time in hours until the patient could successfully achieve this test independently, regardless of the amount of time required.
Time Frame: Hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Control | Experimental
Number analyzed (Participants) | 41 | 39
Hours | 33.4 (7.0) | 46.8 (14.5)

5. Secondary Outcome: Time Until Ambulation at Least 30 Meters
Description: The time in hours until a patient could ambulate at least 30 meters independently (regardless of time to achieve the 30 meters)
Time Frame: 7 postoperative days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Control | Experimental
Number analyzed (Participants) | 41 | 39
Hours | 40.9 (13.0) | 56.6 (16.7)

6. Secondary Outcome: Pain Level
Description: The amount of pain evaluated using the 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Postoperative Days 1-3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 41 | 39
score on a scale
  Postoperative Day 1 (08:00-16:00) | 4.4 (2.0) | 3.7 (2.3)
  Postoperative Day 2 (08:00-16:00) | 3.7 (1.9) | 3.4 (2.1)
  Postoperative Day 3 (00:00-8:00) | 2.5 (2.1) | 2.8 (2.1)

7. Secondary Outcome: Opioid Consumption
Description: Amount of opioid consumed as measured with intravenous morphine equivalents in milligrams
Time Frame: Postoperative Days 0-3
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Control | Experimental
Number analyzed (Participants) | 41 | 39
milligrams
  Recovery Room | 8.6 (7.6) | 8.0 (8.5)
  Postoperative Day 0 (day) | 0.9 (2.3) | 1.5 (4.6)
  Postoperative Day 0 (evening) | 7.2 (6.5) | 8.5 (6.2)
  Postoperative Day 1 (night) | 5.1 (6.7) | 5.6 (6.5)
  Postoperative Day 1 (Day) | 11.0 (6.9) | 12.6 (10.0)
  Postoperative Day 1 (evening) | 8.6 (5.5) | 10.9 (6.3)
  Postoperative Day 2 (night) | 4.1 (4.6) | 5.6 (6.2)
  Postoperative Day 2 (day) | 9.6 (6.5) | 10.2 (6.8)
  Postoperative Day 2 (evening) | 6.5 (5.8) | 7.2 (6.5)
  Postoperative Day 3 (night | 4.9 (6.4) | 5.1 (5.8)

ADVERSE EVENTS:
Time Frame: First postoperative week
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 3/41 | 2/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=41) | Experimental (N=39)
Fall (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) — A fall either from standing or during walking

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No